CLINICAL TRIAL: NCT06404346
Title: Comparative Effectiveness of High Velocity Thrust and Bowen Technique in Patients of SI Joint Dysfunction With Upslipped Innominates. A Randomized Controlled Trial
Brief Title: Comparative Effectiveness of HVT and Bowen Technique in Patients of SI Joint Dysfunction With Upslipped Innominates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/705
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Joint Diseases
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Velocity Thrust (Experimental)
  Interventions: Diagnostic Test: High Velocity Thrust
- Bowen therapy (Other)
  Interventions: Other: Bowen therapy

INTERVENTIONS:
Diagnostic Test: High Velocity Thrust — Group A Participants assigned to the HVT will receive manual therapy sessions consisting of specific manipulative techniques targeting the sacroiliac joint and surrounding structures. participant lying on your side or on your stomach, depending on which SI joint needs to be manipulated.The physiotherapist will stabilize body to isolate the specific SI joint that needs adjustment. This may involve holding certain parts of your body in place or using props like a belt or cushion.With precise control and speed, the physiotherapist will apply a sudden thrust to the targeted SI joint. This thrust aims to mobilize the joint and restore its normal function. This procedure will perform in 3 sessions per week for 2 weeks
  Arms: High Velocity Thrust
Other: Bowen therapy — participants will undergo sessions involving gentle, rolling movements over muscles, tendons, and ligaments in sacroiliac joint . participant lie comfortably on a treatment bed fully clothed, typically face down or on your side. The physiotherapist will perform a series of gentle, rolling movements with their fingers and thumbs over specific points on your body, including the lower back, hips, and buttocks. These moves are designed to stimulate the nervous system and promote relaxation and healing in the affected area.
  Arms: Bowen therapy

SUMMARY:
Sacroiliac joint dysfunction (SIJD) is a common musculoskeletal condition characterized by pain and impaired function in the lower back and pelvis region.

DETAILED DESCRIPTION:
The reported prevalence of sacroiliac joint pain in cases of chronic low back and lower extremity pain is estimated to be between 10 - 27%. Manual therapy techniques, such as High-Velocity Thrust (HVT) and the Bowen Technique, have emerged as potential treatment options for SIJD. HVT involves quick, controlled movements applied to specific joints to restore normal range of motion and alleviate pain. Conversely, the Bowen Technique is a gentle, non-invasive form of bodywork that utilizes subtle rolling movements over muscles and connective tissues to promote relaxation and restore balance within the body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sacroiliac joint dysfunction confirmed by clinical assessment and imaging findings.
* The presence of an upslipped innominate observed on imaging studies.

Exclusion Criteria:

* History of significant trauma or surgery involving the sacroiliac joint region.
* The presence of inflammatory or infectious conditions affecting the sacroiliac joint.
* Contraindications to manual therapy interventions such as HVT or the Bowen Technique.
* Inability to comprehend study procedures or provide informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 12 Months
  used in the management of spinal disorder. The Oswestry Disability Index (ODI) a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.
Visual Analog Scale(VAS) | 12 months
  It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Govt. Hospital Kot Kahwaja Saeed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No